CLINICAL TRIAL: NCT04023734
Title: A Targeted and Tailored Pharmacist Intervention to Improve Adherence to Antihypertensive Drugs Among Patients With Diabetes in Indonesia: a Cluster Randomized Controlled Trial
Brief Title: A Targeted and Tailored Pharmacist Intervention to Improve Adherence to Antihypertensive Drugs Among Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Groningen (Other)
Collaborators: Universitas Padjadjaran (Other)
Responsible Party: Principal Investigator, Sofa Dewi Alfian, Registered pharmacist, University of Groningen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PharIndo2019
Record Dates: First submitted 2019-06-26; First posted 2019-07-17 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension; Medication Nonadherence
Keywords: Medication non-adherence; Type 2 diabetes; Antihypertensive agents
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): A targeted and tailored pharmacist intervention at baseline and at 1-month follow-up.
  Interventions: Behavioral: Reminders, habit-based strategies and/or involvement of family member; Behavioral: Counselling to increase knowledge; Behavioral: Counselling to increase motivation; Behavioral: Explore/address other drug related problems
- Control group (Active Comparator): Usual care based on the Indonesian guideline at baseline and 1-month follow-up.
  Interventions: Behavioral: Usual care based on the Indonesian guideline

INTERVENTIONS:
Behavioral: Reminders, habit-based strategies and/or involvement of family member — Strategies to cope with forgetfulness include reminders, habit-based strategies and/or involvement of family members. The use of a reminder tool and pill boxes will be encouraged and a reminder app can be implemented if patients own a mobile phone. The habit-based strategy will be delivered through a printed worksheet which is tailored to patient's daily routine. Patients will be asked to identify the appropriate place and time to take their medication, and an action they conduct every day that could serve as a prompt or cue to take their medication. Patients will be asked to write coping plans to formulate their own "if-then" plans for all daily doses of their antihypertensive drug(s). Moreover, patients will be asked to choose a family member to become their treatment supporter. This individual will be asked to support patients to take the antihypertensive drugs. Pharmacists will remind patients to take his/her completed worksheet to the next visit.
  Arms: Intervention
Behavioral: Counselling to increase knowledge — The content of the counselling to cope with lack of knowledge will focus on educating patients about the purpose of the medication, when and how to take the medication, the need for long-term use, the importance of medication adherence, and how to deal with possible side effects. To explore which education is needed, the patient will be asked whether they know why and how to take their medication. The teach-back method will be used, where the patient is asked to explain the pharmacist what he/she has understood after receiving the education.
  Arms: Intervention
Behavioral: Counselling to increase motivation — The content of the counselling to cope with lack of motivation will focus on exploring and discussing their concerns and necessity beliefs. This method is called motivational interviewing. This is done by asking a first question about whether the medication bothers the patient. Follow-up on this question can focus on any concerns or low necessity beliefs (e.g., when patients are bothered by the medication because they think the medication is not needed or are afraid of side-effects).
  Arms: Intervention
Behavioral: Explore/address other drug related problems — The content of the counselling to address other drug related problems will focus on exploring these other problems underlying the non-adherence, for example experiencing side effects, costs, polypharmacy, difficulty to refill antihypertensive drugs in time, or medication intake problems, and offering solutions/alternatives when possible.
  Arms: Intervention
Behavioral: Usual care based on the Indonesian guideline — Patients in five CHCs randomized to the control group will receive pharmacist counselling based on the Indonesian guideline of pharmacy practice. At each visit, they will receive information about the quantity and dose of the dispensed drugs, when and how to use and store the drugs, side effects and how to deal with them, the importance of medication adherence, and confirming if the patient understands how to take medications correctly.
  Arms: Control group

SUMMARY:
The primary objective of this study is to assess the effect of a targeted and tailored pharmacist intervention on medication adherence among diabetes patients non-adherent to antihypertensive drugs. The secondary objectives are to assess the effect of the intervention on blood pressure level and medication beliefs, and to evaluate the implementation and adoption of the intervention for pharmacists and patients.

DETAILED DESCRIPTION:
Adherence to chronic medication is often suboptimal. However, existing interventions to improve adherence are either too complex or expensive for implementation and scale-up in low-middle income countries and/or not particularly effective.

A cluster randomized controlled trial with 3-months follow-up will be conducted in 10 Community Health Centers (CHCs) in Indonesia. Patients aged ≥18 years, diagnosed with type 2 diabetes and reported non-adherence to antihypertensive drugs according to the Medication Adherence Report Scale (MARS) are eligible to participate. Patients in the five CHCs randomized to the intervention group will receive a targeted and tailored pharmacist intervention at baseline (first session) and at 1-month follow-up (second session). The intervention will be low-cost, align with the current CHC workflow and will not require a substantial change to the current system. Before dispensing antihypertensive drugs during the first session, the pharmacist will discuss patient-specific barrier(s) for medication adherence based on their responses on MARS and three additional questions, which are derived from the Brief Medication Questionnaires. The intervention strategies will then be tailored to their identified adherence problems. Based on current literature, the investigators defined four non-adherence problems that can be addressed by the community pharmacist, i.e. (1) forgetfulness, (2) lack of knowledge, (3) lack of motivation or (4) other drug-related problems. Of note, patients might need a combined intervention strategy to address all experienced problems. The four non-adherence problems and recommended intervention strategies are specified below:

1. Strategies to cope with forgetfulness include reminders, habit-based strategies and/or involvement of family members.
2. The content of the counselling to cope with lack of knowledge will focus on educating patients about about the purpose of the medication, when and how to take the medication, the need for long-term use, the importance of medication adherence, and how to deal with possible side effects. To explore which education is needed, the patient will be asked whether they know why and how to take their medication. The teach-back method will be used, where the patient is asked to explain the pharmacist what he/she has understood after receiving the education.
3. The content of the counselling to cope with lack of motivation will focus on exploring and discussing the patients' concerns and necessity beliefs (motivational interviewing).
4. The content of the counselling to address other drug related problems will focus on exploring other problems underlying the non-adherence, for example experiencing side effects, costs, polypharmacy, difficulty to refill antihypertensive drugs in time, or medication intake problems, and offering solutions/alternatives when possible.

The follow-up session will be conducted in one month after the baseline session, when patients refill their medication at the next regular outpatient visit. The purpose of the follow-up session is (1) to evaluate the short-term effect of the intervention and discuss the patients' implementation of and experiences with the offered information and recommendations, and (2) to address non-adherence problems that were not yet addressed during the first session. Where needed, the pharmacist, together with patient, can make changes to the coping plan and discuss additional interventions. As the quality of the intervention will depend on the competences and skills of the pharmacist, treatment integrity will be enhanced by an obligatory communication training focusing on motivational interviewing and the teach-back method, and by providing supportive material as part of the intervention.

Patients in five CHCs randomized to the control group will receive pharmacist counselling based on the Indonesian guideline of pharmacy practice. At each visit, they can receive information about the quantity and dose of the dispensed drugs, when and how to use and store the drugs, side effects and how to deal with them, the importance of medication adherence, and confirming if the patient understands how to take medications correctly. Patients in the control group will complete all assessments at the same time points as those in the intervention group

The primary study outcome is the difference between intervention and control group in change in total adherence scores using the MARS between baseline and 3 months follow-up. Secondary outcomes are blood pressure (BP), medication beliefs using the Beliefs about Medicines Questionnaire (BMQ)-specific, and evaluate the intervention using the RE-AIM framework (Reach, Effectiveness, Adoption, Implementation, and Maintenance).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old.
* Diagnosed with type 2 diabetes for at least one year based on patient's medical record.
* Using at least one antihypertensive drug in the last three months.
* Provision of signed informed consent.
* Have sub-optimal medication adherence to antihypertensive drugs according to the MARS (<20).

Exclusion Criteria:

* Patients with severe mental or physical constraints.
* Pregnancy or in the lactation period.
* Illiterate in Indonesian language.
* Enrollment in another intervention study.
* Those not responsible for taking their own medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2019-08-16 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Medication adherence | Baseline, 1-month, and 3-month follow-up
  The differences in change in total score of medication adherence using Medication Adherence Report Scale (MARS). The Indonesian version of the MARS showed to be valid (correlation value of each question to the total score > 0.396) and reliable (Cronbach α coefficient of 0.803). Patients will indicate how often each statement applied to them on a 5-point Likert scale ranging from always (score 1) to never (score 5). Items are summed to obtain a total score ranging from 5 to 25.

SECONDARY OUTCOMES:
Blood pressure level | Baseline, 1-month, and 3-month follow-up
  Within and between patient changes in blood pressure (BP) level (systolic blood pressure [SBP] and diastolic blood pressure [DBP]) at baseline, 1-month, and 3-month follow-up. BP measurements will be performed by a nurse who is blinded to the group assignment.
Medication beliefs | Baseline and 3-month follow-up
  Within patient changes on beliefs about medication will be assessed using the BMQ-specific at baseline and 3-month follow-up. The BMQ-specific contains 5 items about necessity beliefs (e.g. "My health at present depends on my blood pressure-lowering medicines"), and 5 items about concern beliefs (e.g. "I sometimes worry about becoming too dependent on my blood pressure-lowering medicines"). All items have a 5-point Likert scale ranging from strongly disagree to strongly agree with an overall range from 5 (low necessity, low concern) to 25 (high necessity, high concern). A necessity-concern differential score will be calculated by subtracting the scores of the concerns scale from the necessity scale (range -20 to 20). A positive differential score indicates stronger beliefs in the necessity, while a negative score indicates stronger concerns.
Reach | On completion of the final assessments at 3-month follow-up.
  Reach will be assessed by measuring the participation rates and representativeness of patients who participate in this study. In case a patient refuses or discontinues to participate in this study, patient's age, gender, and BP lowering drugs the patient uses will be recorded by research assistants. This information is used to calculate the participation rate and assess differences between responders and non-responders. To determine representativeness, patient's demographics will be compared to census demographics in Bandung City, Indonesia.
Pharmacists' adoption of the intervention | On completion of the final assessments at 1-month follow-up.
  Pharmacists' adoption with various parts of the intervention will be assessed by focus group discussion (FGD). Example of questions:
  * What do you think of the program in general?(Regarding number of sessions, time between sessions, duration of sessions)
  * Tell me about positive experiences you have had with the program. Do others agree? Do others have different experiences?
  * Tell me about negative experiences you have had with the program. Do others agree? Do others have different experiences?
Patients' adoption of the intervention | On completion of the final assessments at 3-month follow-up.
  Patients' adoption with various parts of the intervention will be assessed by a questionnaire (e.g How satisfied are you with the information provided by the pharmacist regarding your antihypertensive drugs during the past three months?)
Pharmacists' suggestions for future implementation | On completion of the final assessments at 1-month follow-up.
  Pharmacists' suggestions for future implementation of the intervention will be assessed by FGD with following questions:
  * Suppose that you were in charge, do you think this program could be implemented in your CHC?
  * Please explain why or why not.
  * What do others think?
  * What do you see as barriers?
  * What would help to support the implementation?
Patients' suggestions for future implementation | On completion of the final assessments at 3-month follow-up.
  Patients' suggestions for future implementation of the intervention will be assessed by a questionnaire (e.g How could we improve the program?)
Pharmacists' willingness to maintain the intervention | On completion of the final assessments at 1-month follow-up.
  Pharmacists' willingness to continue the intervention as part of routine clinical practice over the long term will be assessed by FGD with the following questions:
  * Suppose that this program is implemented, do you think this program will sustain in your CHC? - Please explain why or why not.
  * What do others think?
  * What do you see as barriers?
  * What would help to sustain this program?
Patients' willingness to maintain the intervention | On completion of the final assessments at 3-month follow-up.
  Patients' willingness to continue the intervention as part of routine clinical practice over the long term will be assessed by a questionnaire (e.g Suppose that this program will be implemented in the future, how often would you like to receive it?)

CONTACTS AND LOCATIONS:
Overall Officials: Sofa D Alfian, Principal Investigator — University of Groningen
Locations (1):
- Community Health Centers, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
Other researchers may contact the principal investigator (s.d.alfian@rug.nl)

REFERENCES:
- [Background] Nieuwlaat R, Wilczynski N, Navarro T, Hobson N, Jeffery R, Keepanasseril A, Agoritsas T, Mistry N, Iorio A, Jack S, Sivaramalingam B, Iserman E, Mustafa RA, Jedraszewski D, Cotoi C, Haynes RB. Interventions for enhancing medication adherence. Cochrane Database Syst Rev. 2014 Nov 20;2014(11):CD000011. doi: 10.1002/14651858.CD000011.pub4. PMID 25412402
- [Background] Kini V, Ho PM. Interventions to Improve Medication Adherence: A Review. JAMA. 2018 Dec 18;320(23):2461-2473. doi: 10.1001/jama.2018.19271. PMID 30561486
- [Background] Cutrona SL, Choudhry NK, Fischer MA, Servi AD, Stedman M, Liberman JN, Brennan TA, Shrank WH. Targeting cardiovascular medication adherence interventions. J Am Pharm Assoc (2003). 2012 May-Jun;52(3):381-97. doi: 10.1331/JAPhA.2012.10211. PMID 22618980
- [Background] van Boven JF, Stuurman-Bieze AG, Hiddink EG, Postma MJ, Vegter S. Medication monitoring and optimization: a targeted pharmacist program for effective and cost-effective improvement of chronic therapy adherence. J Manag Care Spec Pharm. 2014 Aug;20(8):786-92. doi: 10.18553/jmcp.2014.20.8.786. PMID 25062071
- [Background] Wroe AL. Intentional and unintentional nonadherence: a study of decision making. J Behav Med. 2002 Aug;25(4):355-72. doi: 10.1023/a:1015866415552. PMID 12136497
- [Background] Clifford S, Barber N, Horne R. Understanding different beliefs held by adherers, unintentional nonadherers, and intentional nonadherers: application of the Necessity-Concerns Framework. J Psychosom Res. 2008 Jan;64(1):41-6. doi: 10.1016/j.jpsychores.2007.05.004. PMID 18157998
- [Derived] Alfian SD, Abdulah R, Denig P, van Boven JFM, Hak E. Targeted and tailored pharmacist-led intervention to improve adherence to antihypertensive drugs among patients with type 2 diabetes in Indonesia: study protocol of a cluster randomised controlled trial. BMJ Open. 2020 Jan 6;10(1):e034507. doi: 10.1136/bmjopen-2019-034507. PMID 31911526